CLINICAL TRIAL: NCT05455775
Title: Video Monitoring FOR Early Signaling of Adverse EvEnts, Technical Validation
Acronym: FORSEE
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Lukas Dekker, Prof. dr. L.R.C. Dekker, Catharina Ziekenhuis Eindhoven
Other Study IDs: CatharinaZE
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Vital Signs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Camera-based monitoring technology — Unobtrusive, vital sign measurement with remote photoplethysmography and laser speckle vibrometry

SUMMARY:
In this study, 30 patients admitted to an high acuity department with hemodynamic or respiratory pathologies will be monitored with camera-based monitoring technologies for 24 hours. The camera's will measure heart rate and respiration rate, based on the principle of remote photoplethysmography and laser speckle vibrometry. Data will be analysed retrospectively and will be compared with vital parameters measured with the standard patient monitor.

DETAILED DESCRIPTION:
Rationale: In hospitals, some 40% of unanticipated deaths occur in low-acuity departments. This alarming figure reflects the limited degree to which the cardiorespiratory status of patients is monitored in these departments, due to the obtrusiveness and expense of existing monitoring technologies, as well as the unpractically high clinical workload and cost that deployment of such technologies would entail.

Objective: This project explores video monitoring of the cardiorespiratory status of the patient as an innovative unobtrusive method that could eventually aid to reduce workload for the staff and better predict (acute) deterioration or adverse cardiac events. The objective of this study is to determine the accuracy and validity of the camera-based vital parameters with respect to the measured contact sensors in intensive care unit (ICU) patients.

Study design: Observational study

Study population: Patients with cardiorespiratory pathologies on the ICU.

Main study parameters/endpoints: The primary end-point is the reliability of the video monitoring technology (remote photoplethysmography and speckle vibrometry) compared with contact sensors focusing on heart rate and respiratory rate in a clinical setting. User experience will have a continuous focus during this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an high acuity unit with a planned stay of at least 4 hours
* Patients with cardiorespiratory pathologies
* Age >= 18

Exclusion Criteria:

* Pregnant patients
* Inability to provide written informed consent
* Mental disability
* Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population within this pilot study will be patients with cardiorespiratory pathologies that are expected to be monitored for at least 4 hours in an high acuity department, which means the Intensive Care Unit, the Medium Care unit or the Coronary Care Unit. This population will be monitored extensively with contact sensors that will serve as the reference to the video-based signals. Most of the patients will recover without any adverse events but some might experience an (acute) cardiorespiratory event (i.e. hemodynamic deterioration).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Validity of the camera-based signals | 24 hours
  Validity of the video based signal compared to the measured signal obtained with a contact sensor.
Feasibility of the camera-based signals | 24 hours
  Feasibility of the video based signal compared to the measured signal obtained with a contact sensor, expressed as percentage of data loss.

SECONDARY OUTCOMES:
Insight in user and patient experience | Within 1 week after intervention
  Insight in user and patient experience with the camera-based monitoring technology

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Dekker, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided